CLINICAL TRIAL: NCT01103102
Title: Phase II Study: Evaluate Dose-Response of Iocide Oral Rinse in a Human Clinical Trial of Gingival Inflammation and Investigate Effects of Biological Markers Indicative of Systemic Disease
Brief Title: Dose-Response Study of Iocide Oral Rinse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20090462H; 1R44HL101821-01 (NIH)
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Gingivitis
Keywords: Gingivitis; Biological Markers
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lowest Dose (Active Comparator)
  Interventions: Drug: Iocide Oral Rinse
- Intermediate Dose (Active Comparator)
  Interventions: Drug: Iocide Oral Rinse
- Highest Dose (Active Comparator)
  Interventions: Drug: Iocide Oral Rinse
- Placebo Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iocide Oral Rinse — Oral Rinse; dosages vary by treatment group; once to twice daily use (depending on treatment group); 12 weeks duration
  Arms: Highest Dose; Intermediate Dose; Lowest Dose
Drug: Placebo — Placebo
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to explore the dose-response relationship of Iocide oral rinse in a clinical trial of gingivitis.

Approximately sixty (60) otherwise healthy subjects having gingivitis will be randomized into the 3-month study to provide 40 total evaluable subjects (10 per group). Each study participant will have four visits: a screening visit up to 21 days before the beginning of the trial, a baseline visit at day 1, and visits at weeks 8 and 12. The duration of the dose/range study will be three months to facilitate compliance and ensure timely completion of the Phase II study.

Three dose/regimens will be evaluated against a placebo control oral rinse. Indices for gingivitis, plaque and bleeding will be scored and blood tests will be performed to determine the effect of the antimicrobial oral rinse on relative levels of biological markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females of at least 18 years of age, and in good general health, as determined by Investigator;
* Have at least 16 natural, gradable teeth and good dental health, as determined by Investigator;
* Have > 25% sites with Gingival Index (GI) scores > 2;
* Have average Plaque Index (PI) score > 2;
* Use of effective method of contraception for the duration of the study or permanently sterilized;
* Able and willing to comply with study requirements including following instructions on study treatment and returning for follow-up visits as required by the protocol;
* Have full understanding of all elements of, and signature and dating of the written informed consent prior to the initiation of protocol specified procedures;
* Females with childbearing potential must have a negative pregnancy test before and during the study period. Sexually active females must be using an effective form of birth control or abstinence. These methods include oral contraceptives ("the pill"), an intrauterine device (IUD), levonogestrel implants (Norplant®), medroxyprogesterone acetate injections (Depo-provera®) or contraceptive foam with a condom.

Exclusion Criteria:

* History, or current evidence, of any significant acute or chronic subject-reported medical or psychiatric condition that, in the opinion of the Investigator, would render examination difficult or invalid or prevent the subject from active study participation;
* ≤24% of sites with GI score >2;
* TPOab positive >34;
* Screening serum level of TSH <0.45 or >4.5;
* Treatment with antibiotic within the one (1) month period prior to the screening examination;
* History of heart murmur, history of rheumatic fever, valvular disease or prosthetic implant requiring antibiotic premedication;
* History of thyroid disease;
* Purported sensitivity or allergy to iodine;
* Known sensitivity or allergy to shellfish;
* History of diabetes;
* History of autoimmune disease;
* Gross oral pathology (periodontal disease, rampant caries, tissue damage created by poor oral care or treatment, soft or hard tissue tumors) that, in the opinion of the Investigator, could influence the outcome of the study;
* Periodontal disease screening will be performed by assessing periodontal pocket depths >5mm on six (6) sites per tooth (distofacial, facial, mesiofacial, mesiolingual, lingual and distolingual). A UNC-15 periodontal probe (Hu-Friedy) will be used for all measurements. Any subject with true periodontal pockets > 5 mm will be excluded from participation in this study;
* Current signs or symptoms of mucosal tissue ulcerations or inflammation, or canker sores;
* Presence of orthodontic appliances or any removable appliance that impinges on the oral tissues being assessed;
* History of early onset periodontal disease or acute necrotizing ulcerative gingivitis;
* Subject reported history in past 6 months or current alcohol abuse that, in the opinion of the Investigator, could influence the outcome of the study;
* Subject reported history of last past 6 months or current drug abuse;
* Use of concomitant medication that, in the opinion of the Investigator, might interfere with the outcome of the study (e.g. antibiotics, immuno-suppressants, steroids, or therapeutic doses of non-steroidal anti-inflammatory agents, phenytoin, calcium antagonists, cyclosporine or coumadin);
* Concomitant therapy with another investigational drug or device without prior approval from the Sponsor within four weeks prior to Visit 2 (Study Day 1);
* Concomitant endodontic or periodontal therapy other than prophylaxis in the past six (6) months;
* Females with childbearing potential with a positive pregnancy test, pregnant or nursing mothers, suspected pregnancy, or intention to become pregnant during the study;
* Residence in the same household as a subject already enrolled in the study (inclusion may create blinding and/or compliance issues);
* Unable and unwilling to comply with the informed consent process, to meet study requirements including following instructions on study intervention, and to return for follow-up visits as required by the protocol;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Gingival Index | Study Day -21 to -7 through Study Day 84
  The primary outcome measure will be the mean gingival index (GI) score.

CONTACTS AND LOCATIONS:
Overall Officials: David L. Cochran, DDS, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States